CLINICAL TRIAL: NCT05633342
Title: Development and Validation of a Blood Test for Screening and Early Detection of Multiple Cancers Based on Circulating Cell-free Nucleic Acid Profiles - Project CADENCE (CAncer Detected Early caN be CurEd)
Brief Title: Project CADENCE (CAncer Detected Early caN be CurEd)
Acronym: CADENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MiRXES Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MX-011-219
Record Dates: First submitted 2022-10-27; First posted 2022-12-01 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Thoracic Cancer; Ovarian Cancer; Liver Cancer; Prostate Cancer; Gastric Cancer; Colorectal Cancer; Breast Cancer; Esophageal Cancer; Pancreatic Cancer
Keywords: MCED; Diagnostic Tests; MiRNA; CfDNA; CtDNA
MeSH Terms: conditions — Ovarian Neoplasms; Liver Neoplasms; Prostatic Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — A total of 30ml of whole blood will be collected in four blood tubes (3 ml in one EDTA tube + 27ml in three Streck Cell-free RNA BCT tubes). Collected blood samples are to be kept at room temperature and processed within 24 hours. All samples are to be processed to obtain separated portions of red blood cells, buffy coat, platelet-rich plasma, and platelet-poor plasma. All samples will be labeled with de-identified subject code and stored at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy average-risk cohort: Individuals representing the general population who self-declare to have no cancer history and have no indications suggestive of underlying cancer development. Subjects will be recruited from a state-of-the-art population study.
- Increased-risk (genetic/familial) cohort: Individuals carrying certain germline mutations that predispose the subjects to an increased risk of having cancer than the general population. Subjects will be recruited from Cancer Genetics Service (CGS).
- High-risk cohort: Individuals diagnosed with diseases that have a high risk of progressing to cancer.
- Malignant cohort: Individuals diagnosed with cancer.

SUMMARY:
With existing evidence showing the difference in miRNA expression levels between non-cancer and cancer groups, the investigators assume that levels of DNA methylation, RNA expression as well as protein concentration will also be dysregulated during disease progression. Combining the power of multi-omic cancer biomarkers, the investigators hypothesize that the sensitivity and specificity of MiRXES MCST can be significantly improved compared to existing multi-cancer diagnostic tests.

In this study, the investigators propose to develop and validate blood-based, multi-cancer screening tests through a multi-omics approach.

DETAILED DESCRIPTION:
This study consists of four (4) objectives:

* Characterize intra-cellular multi-omic profiles of cancer and adjacent normal tissues to aid the selection of circulating cancer biomarkers.
* Select and verify circulating multi-omic cancer biomarkers by characterizing the circulating multi-omic profiles of the peripheral blood of cancer patients, high-risk, increased-risk, and healthy controls, guided by tissue-based cancer omics profiles.
* Develop multi-cancer screening in vitro diagnostic assay(s) based on the selected blood-borne circulating multi-omic cancer biomarker panel(s) and build algorithm(s) to distinguish cancer cases from control groups.
* Clinically validate the performance (AUC, sensitivity, specificity) of the multi-cancer screening assay(s) and algorithm(s)

ELIGIBILITY:
Inclusion Criteria:

Healthy average-risk cohort Individuals representing the general population who self-declare to have no cancer history and have no indications suggestive of underlying cancer development. Subjects will be recruited from a state-of-the-art population study.

Increased-risk (genetic/familial) cohort Individuals carrying certain germline mutations that predispose the subjects to an increased risk of having cancer than the general population. Subjects will be recruited from Cancer Genetics Service (CGS).

High-risk cohort Individuals diagnosed with diseases that have a high risk of progressing to cancer.

Malignant cohort Individuals diagnosed with cancer. Wherever possible, samples for the 'Malignant group' should have a representation of each cancer stage.

Exclusion Criteria:

Pregnant or lactating (self-declaration), unwilling or unable to provide signed informed consent and has or had received chemotherapy or radiotherapy for cancer treatment and/or any other cancer-related treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be carried out in 4 phases, namely Phase 1A, 1B, 1C, and 1D. Phase 1A and 1B will be carried out in parallel. Upon the completion of Phase 1A and 1B, Phase 1C will be initiated, followed by Phase 1D, which is the final phase of this study.
  All four phases involve participant recruitment (except Phase 1A), sample and data collection, and sample data analysis. Subjects recruited for CADENCE will be divided into four groups: (1) Healthy average-risk (2) Increased-risk (3) High-risk and (4) Malignant.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
To discover novel intracellular RNA and methylated DNA cancer biomarkers in fresh frozen tumor tissues. | through study completion, an average of 2.5 years
To select the best-performing multi-omic single-cancer, biomarker panels for each of the cancer types, and develop the corresponding Single-Cancer Early detection Algorithms (SCEAs). | through study completion, an average of 2.5 years
To discover and validate novel cell-free RNA and methylated cell-free DNA cancer biomarkers in the peripheral blood of cancer patients. | through study completion, an average of 2.5 years
To develop the best-performing multi-omic multi-cancer biomarker panel by integration and/or optimization of single-cancer panels and develop the corresponding Multi-Cancer Early detection Algorithm (MCEA). | through study completion, an average of 2.5 years
To develop in vitro diagnostic assay(s) for the Multi-Cancer Screening Test (MCST) and if appropriate Single-Cancer Screening Tests (SCSTs). | through study completion, an average of 2.5 years
To evaluate the clinical performance (AUC, sensitivity, specificity, tissue of origin) of the MCST and if appropriate SCSTs to discriminate cancer cases from control groups. | through study completion, an average of 2.5 years

SECONDARY OUTCOMES:
Secondary outcome: • To explore the relationship between MCST/SCSTs with clinical outcomes based on the collection of longitudinal follow-up information from medical records. | through study completion, an average of 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheng He, PhD, Study Director — MiRXES Pte Ltd
Locations (1):
- Biopollis, Helios, Singapore, Singapore